CLINICAL TRIAL: NCT05974657
Title: Lactobacillus Acidophilus LA85 for Preventing Antibiotic-Associated Diarrhea: A Multi-Centric, Double-Blind, Randomized Study
Brief Title: Effectiveness and Safety of Lactobacillus Acidophilus LA85 in Preventing Antibiotic-Associated Diarrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Collaborators: Methodex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: WK2023001
Record Dates: First submitted 2023-07-07; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Antibiotic Side Effect; Probiotics; Diarrhea
Keywords: diarrhea; probiotics; Antibiotic Side Effect
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): Composition: 400mg maltodextrin (excipient)； Capsule total weight: 400mg； Primary conditioning: HPMC Capsules (Hydroxypropyl Methylcellulose)； Secondary conditioning：Cardboard case Secondary packaging content：14 capsules / blister, 1 blisters per case Dosage regimen: Take one capsule daily before meals； Storage：Store in a cool, dry place without exposure to the sun.
  Interventions: Other: Probiotic Lactobacillus acidophilus LA85
- Probiotic group (Active Comparator): Composition: 20mg (2x109 UFC/ capsule) Lactobacillus acidophilus LA85 (active principle) and 380mg maltodextrin (excipient)； Capsule total weight: 400mg； Primary conditioning: HPMC Capsules (Hydroxypropyl Methylcellulose)； Secondary conditioning：Cardboard case Secondary packaging content：14 capsules / blister, 1 blisters per case Dosage regimen: Take one capsule daily before meals； Storage：Store in a cool, dry place without exposure to the sun.
  Interventions: Other: Probiotic Lactobacillus acidophilus LA85

INTERVENTIONS:
Other: Probiotic Lactobacillus acidophilus LA85 — Through a randomized double-blind placebo-controlled method, the patients were randomly divided into placebo group and probiotic intervention group, and took probiotics once a day for 14 consecutive days.

SUMMARY:
This randomized, placebo-controlled, double-blind clinical trial aims to evaluate the efficacy and safety of probiotics as food supplements in preventing antibiotic-associated diarrhea. The study will involve 82 patients who will be randomly assigned to one of two groups: an experimental group receiving a probiotic containing Lactobacillus acidophilus LA85, and a placebo group. The primary outcomes measured include the number of days until the onset of diarrhea, the duration of diarrhea (if it occurs), gastrointestinal quality of life evaluation using the GIQLI questionnaire, and overall patient satisfaction.

DETAILED DESCRIPTION:
This randomized, placebo-controlled, double-blind clinical trial aims to assess the effectiveness and safety of probiotics as food supplements in preventing antibiotic-associated diarrhea. The study will enroll 82 patients who will be randomly assigned to either the experimental group or the placebo group. Participants in the experimental group will receive a probiotic supplement containing Lactobacillus acidophilus LA85, while those in the placebo group will receive a non-active substitute.

The outcomes include the following measurements:

1. Number of days until the onset of diarrhea.
2. Duration of diarrhea, if it occurs.
3. Evaluation of gastrointestinal quality of life using the GIQLI questionnaire.
4. Overall patient satisfaction with the intervention. Throughout the trial, a double-blind approach will be maintained, ensuring that both the participants and the investigators are unaware of the treatment assignments. This helps minimize bias and ensures the reliability of the results. To assess the efficacy and safety of probiotics, data will be collected and analyzed using appropriate statistical methods. The number of days until the onset of diarrhea will be compared between the two groups, as well as the duration of diarrhea if it occurs. Gastrointestinal quality of life will be evaluated using the GIQLI questionnaire, which measures various aspects related to gastrointestinal well-being. Additionally, overall patient satisfaction with the intervention will be assessed. By conducting this comprehensive clinical trial, we aim to provide valuable insights into the potential benefits and safety of probiotics as food supplements in preventing antibiotic-associated diarrhea. The results obtained will contribute to evidence-based recommendations for healthcare professionals and may have implications for improving patient outcomes and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients starting antibiotic treatment (Amoxicillin 750mg).
* Patients prone to diarrhea with the administration of Amoxicillin 750mg.
* Patients over 18 years of age.
* Patients of both sexes.
* Patients capable of understanding the clinical study and who are committed to complying with the requirements and procedures of the study.
* Patients who have signed the informed consent.

Exclusion Criteria:

* Diabetic patients.
* Pregnant patients.
* Patients who are breastfeeding.
* Patients who require pharmacological treatment that triggers drug diarrhea (laxatives, antacids with magnesium, chemotherapy, omeprazole, esomeprazole, lansoprazole, rabeprazole, cimetidine ranitidine, mycophenolate nizatidine, ibuprofen, naproxen and metformin).
* Patients requiring treatment with tricyclic antidepressants, antiepileptics, antihistamines, antiparkinsons, antipsychotics, antispasmodics, verapamil, monoamine oxidase inhibitors, opiates, sympathomimetics, antacids (with aluminum and calcium), non-steroidal antidiarrheals and anti-inflammatory drugs.
* Patients who change the type of diet during the study.
* Patients with an allergy or intolerance to any of the ingredients in the formulation of the product under study.
* Subjects with a history of drug, alcohol or other substance abuse, or other factors that limit their ability to cooperate during the study.
* Subjects whose condition does not make them eligible for the study, according to the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Diarrhea Onset Time | 14 days
  Evaluate stool characteristics on the Bristol Scale (Degree 5-7 indicative of diarrhea).

CONTACTS AND LOCATIONS:
Overall Officials: Joan Ciurana, Dr., Principal Investigator — Dentist Ciurana Clinic; Xavier Calvo, Dr., Principal Investigator — Dentist Rob Clinic
Locations (1):
- Ciurana Clinic, Barcelona, Castelldefels, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu J, Sun Y, Dong Y, Zhao Y, Gai Z, Fang S. Efficacy and Safety of Lactobacillus acidophilus LA85 in Preventing Antibiotic-Associated Diarrhea: A Randomized, Placebo-Controlled Study. Food Sci Nutr. 2025 Jun 20;13(6):e70490. doi: 10.1002/fsn3.70490. eCollection 2025 Jun. PMID 40548185